CLINICAL TRIAL: NCT04305002
Title: Effect of Exenatide on Disease Progression in Early Parkinson's Disease
Brief Title: Exenatide Treatment in Parkinson's Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Center for Neurology, Stockholm (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Per Svenningsson, MD, Professor, Center for Neurology, Stockholm
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ExPD-ESR-18-13512
Record Dates: First submitted 2020-02-20; First posted 2020-03-12 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Parkinson Disease
Keywords: Glucagon-Like Peptide 1; Positron-Emission Tomography
MeSH Terms: conditions — Parkinson Disease | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Exenatide (Experimental)
  Interventions: Drug: Exenatide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Exenatide — Injections, 2 mg once weekly for 18 months
  Arms: Exenatide
Drug: Placebo — Injections, once weekly for 18 months
  Arms: Placebo

SUMMARY:
The development of a disease-modifying therapy that delays, reverses or stops the symptom progression remains the most important unmet goal in the treatment of Parkinson's disease (PD). Apart from its glucose lowering effect, glucagon-like peptide-1 (GLP-1) receptor stimulation has been investigated in animal models of PD and shown to increase neurogenesis, to arrest and possible reverse nigrostriatal damage, and to protect dopaminergic neurons from neurodegeneration. Exenatide is a synthetic analogue of human GLP-1, resistant to the metabolic processes that degrade it in its naturally occurring form. Results from a recent randomised, double-blind, placebo-controlled trial in PD showed that patients in active treatment for one year were improved compared to the placebo arm with regard to their performance in Movement Disorders Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) motor subscale in the practically defined OFF medication state.

The aim of this trial is to investigate the effect of Exenatide, 2 mg, subcutaneous injection, once weekly on disease progression represented by the change in longitudinal Positron emission tomography with 2-deoxy-2-[fluorine-18]fluoro- D-glucose (FDG-PET) in individual PD subjects, and to identify an Exenatide-related pattern in FDG-PET that will provide insight into the treatment-effect in the brain. The investigators chose the standard regimen prescribed in Type 2 Diabetes Mellitus (T2DM) and the regimen used in a recent trial in PD. The treatment period will be 18 months, and patients will be randomly assigned to either active treatment or placebo. Patients with PD diagnosis, stable on medication during the last year, and Hoehn and Yahr stage 2 or less will be evaluated for the inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of clinically probable Parkinson's disease according to the MDS clinical diagnostic criteria for PD
* Males or Females
* Hoehn and Yahr stage ≤ 2 in the ON medication state. This implies that all patients will be mobile without assistance during their best "ON" medication periods.
* Patients are on levodopa treatment.
* No need for extended treatment adjustment, no significant motor fluctuations during the last year.
* All patients will be ≥25 and ≤80 years of age
* Ability to self-administer, or to arrange carer administration of the trial drug.
* Signed informed consent to participate in the trial.

Exclusion Criteria:

* Atypical or other causes of parkinsonism. Patients with suspected Multiple System Atrophy, Progressive Supranuclear Palsy, drug-induced parkinsonism, vascular parkinsonism, dystonic or essential tremor will not be included in the trial.
* Prior intra-cerebral surgical intervention for Parkinson's disease. Patients who have previously undergone Deep Brain Stimulation, intra-cerebral administration of growth factors, gene therapy or cell therapies will not be eligible.
* Already actively participating in a trial of a device, drug or surgical treatment for Parkinson's disease.
* Previous exposure to Exenatide.
* Known abnormality on CT or MRI brain imaging considered likely to compromise compliance with trial protocol/FDG-PET acquisition.
* Patients with body mass index below 18.5. Exenatide causes weight loss, and individuals with already low BMI will not be eligible.
* Patients with diabetes mellitus type 1.
* Patients with prediabetes (HbA1c at screening 42-47 mmol/mol), or T2DM (known diagnosis, ongoing antidiabetic treatment or HbA1c > 47 mmol-mol and fasting plasma glucose > 7.0 mmol/L at screening).
* History of pancreatitis. Baseline serum amylase value should be within the laboratory normal range +/- 20 percent.
* Severe gastrointestinal disease including gastroparesis.
* History of alcoholism.
* History of severe cardiac disease.
* History of pancreas cancer.
* History or suspicion of thyroid cancer. Undiagnosed neck lump, hoarse voice, or difficulty swallowing not attributable to PD.
* Personal or family history of medullary thyroid cancer.
* Patients with Multiple Endocrine Neoplasia 2 (MEN2) syndrome.
* End stage renal disease or creatinine clearance < 50 ml/min.
* Hyperlipidaemia. A lipid profile will be tested at the screening visit. Cholesterol or Triglyceride levels greater than 2 x the upper limit of normal will raise suspicion of a familial or acquired hyperlipidaemia and will prompt referral to a relevant specialist for investigation and treatment.
* Concurrent treatment with warfarin.
* Concurrent severe depression, defined as MADRS score 16.
* Concurrent dementia, defined as Mini-Mental State Examination (MMSE) < 22.
* Pregnancy and Breastfeeding.
* There are no safety data regarding Exenatide use in pregnancy. Women of childbearing potential should only be included after a confirmed menstrual period and a negative highly sensitive urine or serum pregnancy test, and will be asked at each visit to confirm regular use of an effective method of contraception. Those who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and until the end of the relevant systemic exposure period (i.e. 10 weeks after the last dose of study drug) will not be eligible. The following birth control methods are considered to be acceptable: combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal or transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, intravaginal or transdermal), intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomised partner, and sexual abstinence.
* Known hypersensitivity or allergy or intolerance to GLP-1.
* Known hypersensitivity to Exenatide or any of its excipients.
* Potential participants who lack the capacity to give informed consent
* Any medical, psychiatric or other condition which in the investigator's opinion compromises the potential participant's ability to participate in the trial.

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2023-10-10 (Estimated); Study Completion 2023-10-10 (Estimated)

PRIMARY OUTCOMES:
FDG-PET network analysis | 21 months

SECONDARY OUTCOMES:
The sum score of MDS-UPDRS part 3 in ON and OFF-medication state | 18 and 21 months
MDS-UPDRS part 2 | 9, 18 and 21 months
MDS-UPDRS part 4 | 9, 18 and 21 months
Hoehn and Yahr | 18 and 21 months
Accelerometer (intensity of physical activity) | 18 and 21 months
Accelerometer (steps per day) | 18 and 21 months
Accelerometer (time of inactivity per day) | 9, 18 and 21 months
Levodopa equivalent daily dose (LEDD) | Every 3 months
PDQ-39 mobility subscore | 18 months
MDS-UPDRS part 1 | 18 and 21 months
  Non-motor symptom progression
Non-Motor Symptoms Questionnaire (NMSQuest) | 18 months
  Non-motor symptom progression
PDQ-39 subscores (except for mobility) | 18 months
  Non-motor symptom progression
Epworth Sleepiness Scale (ESS) | 18 months
  Non-motor symptom progression
MADRS | 6, 12 and 18 months
  Non-motor symptom progression
Montreal Cognitive Assessment (MoCA) | 21 months
  Non-motor symptom progression
Brief Smell Identification Test (B-SIT) | 18 months
  Non-motor symptom progression
Frequency and severity of Adverse Events | 21 months
Exenatide-concentration csf | Baseline, 9 and 21 months
Exenatide levels in serum | Baseline, 9, 18 and 21 months

CONTACTS AND LOCATIONS:
Overall Officials: Per Svenningsson, Principal Investigator — Academic Specialist Center, Center for Neurology, SLSO
Locations (1):
- Academic Specialist Center, Center for Neurology, SLSO, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided